CLINICAL TRIAL: NCT07208825
Title: The Effectiveness of Individualized Physical Therapy and Functional Neurology Treatment Protocol in Conjunction With Optimizing Medication and Repetitive Transcranical Magnetic Stimulation in Patients With Complex Regional Pain Syndrome.
Brief Title: The Effectiveness of Conservative Treatment in Patients With Complex Regional Pain Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Collaborators: The Maud Kuistila Memorial Foundation (Unknown)
Responsible Party: Principal Investigator, Jani Takatalo, Associate Chief Physician, Pain Clinic, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EETTMK: 6/2024
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: CRPS (Complex Regional Pain Syndromes)
Keywords: CRPS; GMI; Graded motor imaginary; Rehabilitation; Functional neurology; rTMS; medication
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Some care providers (rTMS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (Active Comparator): Optimizing medication (6mo) followed by rTMS and basic physical therapy rehabilitation (6mo)
  Interventions: Device: rTMS; Other: Basic physical therapy treatment; Other: Functional neurology; Drug: Optimizing the medication
- Early functional neurological rehabilitation (Experimental): Early functional neurological rehabilitation with optimizing medication (6mo) followed by rTMS and basic physical therapy rehabilitation (6mo)
  Interventions: Device: rTMS; Other: Basic physical therapy treatment; Other: Functional neurology; Drug: Optimizing the medication
- Early maximal rehabilitation (Experimental): Early functional neurological and physical therapy rehabilitation with optimizing medication (6mo) followed by rTMS (6mo)
  Interventions: Device: rTMS; Other: Basic physical therapy treatment; Drug: Optimizing the medication
- Basic treatment protocol (Other): Early physical therapy rehabilitation with optimizing medication (6mo) followed by rTMS (6mo)
  Interventions: Device: rTMS; Other: Basic physical therapy treatment; Drug: Optimizing the medication

INTERVENTIONS:
Device: rTMS — 2 weeks starting period (10 treatment days) followed by 5 treatment once a month.
Other: Basic physical therapy treatment — 10 sessions with physical (or occupational) therapist with special education for treating CRPS
Other: Functional neurology — 4 to 6 sessions with specialized OMT-physical therapist who will aim to improve the neurological deficits of the CRPS patient
  Arms: Control group; Early functional neurological rehabilitation
Drug: Optimizing the medication — Aim is to optimize the medication of the CRPS patient according the the medication guidelines

SUMMARY:
The aim of the study is to investigate and improve non-pharmacological rehabilitation methods for patients with Complex Regional Pain Syndrome (CRPS) to reduce pain and restore work and functional capacity to lower overall treatment costs. Current treatment methods offer limited rehabilitation potential for this challenging pain condition, so efforts should be made to raise the level of care and rehabilitation for a disease that often causes long-term and severe reductions in patients' functional and occupational abilities. CRPS patients almost always have to substantially reduce their work hours or withdrawn from the workforce for extended periods, and often permanently, increasing the urgency of strengthening rehabilitation approaches; a CRPS symptoms can end a patient's productivity for society. In addition, commonly used medications are a significant expense for both individuals and the healthcare system. CRPS rarely resolves fully, and even with extensive rehabilitation only a small proportion of patients regain sufficient improvement to return to work at a level of at least 60% capacity.

Participants will be recruited from the Department of Physical Medicine and Rehabilitation at Oulu University Hospital, where CRPS diagnostics for the Northern Ostrobothnia area are primarily conducted. The study will be carried out at OYS rehabilitation outpatient clinics. A total of 39 participants will be recruited into each of four study groups, for an overall sample size of 156 individuals. Each study group will receive repetitive transcranial magnetic stimulation (rTMS) at some point, and functional neurological rehabilitation will be combined with rTMS in varying ways (content and timing will differ between groups). All participants will receive basic CRPS rehabilitation (physiotherapy and occupational therapy) that is provided for all RPS patients, and the timing of this relative to rTMS will also be varied. Recruitment is planned to begin in a autumn 2025.

DETAILED DESCRIPTION:
Complex Regional Pain Syndrome (CRPS) is a disabling and painful pain syndrome. It can be triggered by a very minor injury or a routine surgery, and the symptoms last much longer and are more difficult than the normal healing process would suggest. Symptoms of CRPS can include sensory and motor disorders, autonomic disorders, functional deficits, and major challenges in coping with daily activities. In addition, patients often have challenges with sleeping. Therefore, a multidisciplinary approach is required for treatment, even for several years. Treatment options include medication, rehabilitation (physiotherapy and occupational therapy), psychological interventions, surgical interventions, and alternative therapies. The best evidence currently exists for mirror therapy and Graded Motor Imaginery (GMI)-type rehabilitation interventions, although the evidence for these is based on a relatively small number of original studies. A new form of rehabilitation has emerged as functional neurological rehabilitation, which aims to optimize the functioning of the nervous system and thereby improve the symptoms and functional capacity of CRPS patients. This approach has not yet been extensively studied in CRPS patients.

Magnetic stimulation therapy (repetitive transcranial magnetic stimulation, rTMS) has been used effectively to treat many types of pain conditions (neuropathic pain, musculoskeletal pain, etc.) since the early 2000s. In rTMS therapy, a magnetic field is generated in the head area using an electromagnetic coil, which can affect the excitability level of the nerves in the stimulated area, but also in areas outside the magnetic field through extensive nerve connections. rTMS therapy can irritate or calm the excitability threshold of the nerves. There are also some studies conducted with a small sample size on the treatment of CRPS using rTMS with relatively good results. The effectiveness of the treatment seems to emerge with a slight delay. However, in a recent meta-analysis and recommendations for the use of rTMS therapy, the treatment is recommended for CRPS patients. (Chang et al 2020, Lefaucheur et al 2020.) The aim of the study is to investigate the significance of the timing of CRPS rehabilitation and functional neurological rehabilitation implemented at OYS in relation to rTMS treatment in alleviating symptoms and improving functional capacity in CRPS patients. The aim is also to monitor the effectiveness of the patients' treatment over a long period of time (1 and 3 years).

Study population and research methods The study population consists of patients from the OYS physiatry (or pain clinic) who have been referred for assessment from primary health care or other OYS clinics to make or confirm a CRPS diagnosis. After a CRPS diagnosis is made, the patient's possible initiation of rTMS treatment is discussed in a multidisciplinary pain working group. Patients for whom rTMS treatment is considered a suitable form of treatment will be asked about their willingness to participate in a treatment study for CRPS patients. The inclusion criteria are patients aged 18-70 who can understand Finnish fluently (reading and speaking) and who voluntarily participate in the study. In addition, the patient's CRPS symptom must be in 1-3 limbs. CRPS that has spread to the body or more than 3 limbs is an exclusion criterion. The patient's CRPS must also have developed within less than 5 years, even if the diagnosis is only made during the initial assessment by the OYS physiatrist, i.e. CRPS patients over 5 years old are excluded from the study.

All those receiving rTMS treatment who understand Finnish will be connected to the rTMS digital treatment pathway, which will allow their situation and symptoms and the effectiveness of the treatment to be monitored as part of the clinical work. Before the start of rTMS treatment, a magnetic resonance imaging (MRI) of the head will be taken from the patient to plan the treatment, as the treatment area(s) will be planned using this individual "brain map". The standard rTMS treatment protocol includes a 2-week intensive treatment period (5 + 5 days) and then maintenance treatments once a month for 5 times, i.e. the total treatment period is 6 months. If necessary, the patient is contacted by phone. As long as the patient is on rTMS treatment, he or she is followed up on the digital treatment path and the patient's situation is also inquired about 3 and 6 months after the end of treatment via the digital treatment path. The material collected on the digital treatment path is used as part of the study data collection from the patients participating in the study. The digital treatment path has been implemented and all rTMS treatments are connected to the digital treatment path. There are several surveys on the digital treatment path which include the following:

Before the start of the rTMS treatment period: Jenkins sleep questionnaire, Beck Depression Inventory, quality of life questionnaire, visual analogue scale (pain questionnaire), amount of sleep and changes in well-being.

Patients entering the study will complete an informed consent form, after which they will be randomly assigned to one of four treatment groups. The randomization will be done in groups of 12 people, so that the different groups will have an even distribution of subjects throughout the study. The four treatment groups are:

1. Group 1: Late initial rehabilitation and rTMS; CRPS initial rehabilitation (occupational and physiotherapy according to individual needs, approximately 10 outpatient visits) and rTMS treatment simultaneously after optimization of drug treatment simultaneously.
2. Group 2: Neurological rehabilitation and rTMS; Neurologically focused initial rehabilitation group before the start of rTMS treatment and initial rehabilitation according to the normal treatment protocol.
3. Group 3: Enhanced initial rehabilitation and late rTMS; CRPS initial rehabilitation and functional neurological rehabilitation initially and then rTMS treatment
4. Group 4: OYS's so-called normal treatment; CRPS initial rehabilitation followed by rTMS treatment according to the current normal treatment protocol.

All study groups will receive OYS's minimum rehabilitation aimed at CRPS patients, but one treatment group will only receive initial rehabilitation at the same time as drug treatment optimization and rTMS treatment. All participants in the study will receive a period of rTMS treatment. Before randomization to groups, the severity of the patients' CRPS will be assessed using a dedicated scale. For a large proportion of CRPS patients, an rTMS treatment period is planned at the OYS unless there are contraindications to the treatment or previous examinations (head MRI). For all groups, drug treatment optimization will be implemented during the first 6 months of diagnosis.

The treatment of study group 1 includes drug treatment optimization during the first 6 months and then CRPS initial rehabilitation and rTMS treatment will be implemented simultaneously. rTMS treatment (6 months including a maximum of 15 treatment sessions) and CRPS initial rehabilitation (approx. 10 times) then begins at 6 months. CRPS initial rehabilitation includes a maximum of 10 treatment sessions together with a physiotherapist and/or occupational therapist, some of the appointments are joint appointments. Exercises and rehabilitation progress are selected individually. Initial rehabilitation includes the following areas and their emphasis areas are selected individually: assessment of rehabilitation goals, two-point discrimination, sleep guidance, relaxation training, GMI (including mirror therapy), balancing rest and activity (pacing), pressure garment assessment, therapeutic exercises, making activity/exercise plans, pain experience meter and hardening treatment. Initial rehabilitation usually lasts approx. 6 months.

In study group 2, the practice of functional neurology begins immediately after the CRPS diagnosis is made. rTMS treatment and CRPS initial rehabilitation (approx. 10x) then begin at 6 months at the latest. Functional neurological rehabilitation includes optimizing the neurophysiology of movement and pain and the cooperation of cranial nerves to improve brain plasticity, reduce the threat state experienced in the brain by inhibiting and activating specific nerve connections with individual exercises and thereby relieve pain. There are a total of 4-6 treatment sessions per subject at 3-6 week intervals, i.e. the functional neurology treatment period is carried out before the start of rTMS treatment. The first functional neurology rehabilitation visit is 90min (+ 30min recording time) and the following visits are 45min (+ 15min recording time).

In research group 3, CRPS initial rehabilitation and functional neurological are carried out during the first 6 months, and then an rTMS treatment period is carried out.

In research group 4, the starting point is the current rehabilitation of the OYS, i.e. initial rehabilitation is carried out during the first 6 months, and then an rTMS treatment period is carried out. The groups and schedule are shown in Figure 1 (flow-chart).

The number of subjects has been calculated with two main variables, pain and patient-specific functional scale (PTA), Taking into account a possible 20% dropout rate, the total number will be 156, i.e. 39 subjects in each group. The study will start in autumn 2025.

A multidisciplinary rehabilitation team (physician, physiotherapist, occupational therapist and pain psychologist) will implement the rehabilitation of CRPS patients at OYS. Patients are selected for rTMS treatment by a multidisciplinary pain working group, which includes all healthcare professionals from the pain clinic and, for example, representation from clinical neurophysiology and psychiatry. This working group assesses patients who would potentially benefit from rTMS treatment and assesses whether the patient has any potential contraindications to the treatment or to MRI imaging of the head. In addition, the doctor who diagnosed the patient with CRPS at the physiatry clinic will also review any potential contraindications to treatment and imaging. There are no actual contraindications to rehabilitation and functional neurological rehabilitation. The patient must be able to commit to the exercises they receive from the rehabilitation.

The initial assessment is carried out at the physiatry outpatient clinic at the doctor's office, where a CRPS diagnosis is made and its severity is assessed. Basic data can be collected from all subjects via the digital path, so there is no need to order large numbers of additional surveys. In initial rehabilitation, an initial assessment is carried out by an occupational and physiotherapist. The same therapists make the same assessments again at the end of the initial rehabilitation (see the indicators section). Physiotherapists and occupational therapists are physiotherapists working at the physiatry outpatient clinic who have long-term experience in the rehabilitation of CRPS patients. The rehabilitation is a normal outpatient activity.

rTMS treatments are also carried out as normal outpatient activities in the clinical neurophysiology and physiatry clinics to the extent that equipment and staff capacity allow. rTMS treatments are carried out by a nurse who has received additional training in administering rTMS treatments as normal work at the KNF clinic. The MRI scans of the head are carried out according to the normal protocol. Functional neurological rehabilitation is only just beginning to spread from the world to Finland, and in this regard, there is only one expert in this field in Finland (OMT physiotherapist).

All those involved in the study are healthcare professionals and are subject to a confidentiality obligation. The patient's information is encoded under a numerical study code everywhere when transferring patient data outside the patient information system (SPSS, Excel) and only the people doing the administrative work of the study can access this information, as this information is behind password-protected storage systems.

Measures The main measures of the study are the patient-specific functional scale (PTA) and the pain questionnaire (VAS). In addition, patients will be measured on the rTMS digital therapy path for sleep quality (Jenkins sleep questionnaire), sleep quantity (open question), mood (BDI; Beck Depression Inventory), fear-avoidance behavior (FABQ; Fear-Avoidance Beliefs Questionnaire), mood (DEPS), self-efficacy (PSEQ; Pain Self-Efficacy Questionnaire), quality of life (15D), changes in well-being (open-ended question), fear of movement (TSK; Tampa Scale of Kinesiophobia), left-right discrimination of the symptomatic limb and two-point discrimination ability at the beginning of the study, at 6 months and at 1 year. At these three time points, thermal imaging of the CRPS limb will also be performed. In addition, the patient's medications and condition can be monitored during the study from patient document notes and via the rTMS digital treatment path.

It is not possible to blind the subjects or therapists to the therapies being implemented in the study, but it is possible to blind the persons providing the treatments to some of the measurement results (especially the person implementing the functional neurological rehabilitation).

ELIGIBILITY:
Inclusion Criteria:

* CRPS symptoms maximum of 5 year at the time of diagnosis (CRPS 1 and 2)
* 18 to 70-year-old
* rTMS treatment is granted by university hospital pain clinic (by multidisciplinary group)
* Voluntary to participate into the study

Exclusion Criteria:

* CRPS symptoms started over five years ago (although diagnosed first time now)
* No other outpatient/inpatient rehabilitation during the study rehabilitation period (insurance company or other third party)
* Under 18-years-old of over 70-years-old
* No eligible to rTMS treatment or for other reason rTMS treatment was not granted by university hospital pain clinic (by multidisciplinary group)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient specific functional scale (PSFS) | Enrollment, 6, 12 and 36 months.
  Patient names three important tasks that are compromised by the CRPS and label them by number (from 0 to 10) according the to the ability to perform them at the day of evaluation. Higher the number, better the function (from 0 to 30)
Visual analog scale (VAS) | Enrollment, 6, 12 and 36 months
  Participant is asked to mark with a vertical line the pain experienced during the day of evaluation into the 10cm horizontal line.

SECONDARY OUTCOMES:
Jenkis sleep questionnaire | Enrollment, 6, 12 and 36 months. During the rTMS treatment
  a four-item self-report instrument designed to efficiently screen for the frequency and intensity of common sleep disturbances
Amount of sleep | Enrollment, 6, 12 and 36 months. During the rTMS treatment
  Open question on average hours of sleep during the last week
Beck Depression Inventory | Enrollment, 6, 12 and 36 months
  a 21-item, self-report questionnaire designed to screen for and measure the severity of depression in adults and adolescents
DEPS | Enrollment, 6, 12 and 36 months
  10 item depression questionnaire
Pain Self-Efficacy Questionnaire (PSEQ) | Enrollment, 6, 12 and 36 months
  a 10-item questionnaire developed to assess the confidence people with ongoing pain have in performing activities while in pain
15D | Enrollment, 6, 12 and 36 months
  A generic, comprehensive (15-dimensional), self-administered instrument for measuring Health Related Quality of Life among adults

OTHER OUTCOMES:
General well-being question | ENrollment, 6, 12 and 36 months
  Open question
Tampa Scale of Kinesiophobia | Enrollment, 6, 12 and 36 months
  a 17-item self-report questionnaire designed to measure fear of movement or re-injury, particularly in patients with chronic pain
Right-left discrimination | Enrollment, 6, 12 months
  the ability to differentiate between the left and right sides of one's body and the external world (test is performed with iPad)
Two-point discrimination | Enrollment, 6, 12 months
  a neurological assessment of tactile spatial acuity, measuring the ability to perceive two simultaneous points of touch as separate rather than one (affected and non-affected limb)

CONTACTS AND LOCATIONS:
Overall Officials: Jani M Takatalo, PhD, MD, PRM Specialist, Principal Investigator — Oulu University Hospital, Pain Clinic
Locations (1):
- Oulu University Hospital, Pain Clinic, Oulu, North Ostrobothnia, Finland

IPD SHARING:
Plan to Share IPD: Undecided
This is not decided yet